CLINICAL TRIAL: NCT04379609
Title: Masticatory Efficiency Before and After Muscle-Related Temporomandibular Disorder Treatment
Brief Title: Effects of Temporomandibular Disorder on Masticatory Efficiency
Status: Completed | Type: Observational
Sponsor: Bahçeşehir University (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ezgi Yüceer Çetiner, Assistant Professor, Bahçeşehir University
Other Study IDs: 2017/410
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Temporomandibular Disorder
Keywords: chewing efficiency; masticatory efficiency; masticatory muscles; masticatory performance; temporomandibular disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Employees and students: The control group was selected from among the employees and students of the faculty of dentistry to represent the general population without any temporomandibular disorder (TMD).
  Interventions: Other: Masticatory efficiency
- Patients: Patients who were referred to the Ondokuz Mayıs University Faculty of Dentistry Department of Prosthodontics with a complaint of pain in the chewing muscles were enrolled in this study.
  Interventions: Other: Masticatory efficiency

INTERVENTIONS:
Other: Masticatory efficiency — Two-color chewing gum mixing ability test was used to measure masticatory efficiency in the control group, before and after treatment in the experimental group.21 Commercial two-color chewing gum was used.The gum was left on the patient's tongue and he/she was asked to chew 20 times naturally.
  After chewing, the gum was put in a transparent plastic bag and squeezed to 1 mm. Both sides of the sample were scanned at 300 dpi resolution on a desktop scanner (HP Deskjet, California, USA) in the same day to prevent the colors from deteriorating due to saliva. For each patient, two sides of scanned images were processed in ViewGum software (version 1.4, Dhal Software, Kifissia, Greece, www.dhal.com) using the method of Halozenitis et al. (2013).22 The value of VOH (variance of hue) was taken as the value of chewing activity. The highness of this value indicates low masticatory efficiency.

SUMMARY:
Temporomandibular disorders (TMD) are defined by pain in the temporomandibular joint (TMJ) and related tissues, limitations in the movements of the lower jaw, and TMJ noises.1,2 TMD are classified into four groups as temporomandibular joint disorders, masticatory muscle disorders, headache attributed to TMD and associated structures.3,4 Of these, masticatory muscle disorders are the most common TMD subtype seen in dental clinics.5-7 In general, two major symptoms are seen associated with masticatory muscle disorders: Pain and dysfunction. Pain is the vast majority of complaints about masticatory muscle disorders. The other important complaint is dysfunction, which occurs as a limitation in the opening range of the mandible.8 It is known that individuals with experimental muscle pain are slower than healthy individuals when biting hard food and show lower maximum voluntary clenching capacity.9 Also, it has been reported that the maximum bite force decreased in patients with temporomandibular disorders.10 These consequences directly affect patients' quality of life. Therefore, rehabilitation of limited masticatory functions is one of the important therapeutic goals for TMD patients.11 In TMD patients, masticatory functions can be measured objectively with bite force, bite force endurance, electromyography, and jaw kinematics, etc. Another objective method that can be used to determine masticatory functions is the masticatory efficiency test. In the literature, there are few studies that measure masticatory efficiency in TMD patients.12-16 Only two of these studies investigated the effect of TMD treatment and used the sieve method to measure masticatory efficiency.15,16 Although the sieve method is considered the gold standard, the procedure is complex and time consuming.17,18 To eliminate these disadvantages, masticatory efficiency measurement with two-color chewing gum tests which are simple and do not require special equipment or training can be used. The effect of many different conditions and treatments on masticatory efficiency was evaluated with this method.19 However, to our knowledge, there is no study in the literature evaluating TMD treatment with this method.

The aim of this study was to compare the masticatory efficiency with a two-color chewing gum test before and after treatment of the masticatory muscle-related temporomandibular disorder.

ELIGIBILITY:
Inclusion Criteria:

Presence of muscle-related temporomandibular disorder

Exclusion Criteria:

Patients under the age of 18, who had a missing tooth (except 3rd molars) or crown-bridge restorations, any intra-articular temporomandibular disorder were excluded from the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 21 patients who were referred to the Ondokuz Mayıs University Faculty of Dentistry Department of Prosthodontics with a complaint of pain in the chewing muscles were enrolled in this study. The control group was selected from among the employees and students of the faculty of dentistry to represent the general population without any temporomandibular disorder (TMD).
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-11-03 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
masticatory efficiency | 6 weeks
  Two-color chewing gum mixing ability test was used to measure masticatory efficiency in the control group and experimental group

CONTACTS AND LOCATIONS:
Locations (1):
- Ezgi Yüceer Çetiner, Istanbul, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No